CLINICAL TRIAL: NCT01067755
Title: Clinical Product Evaluation of the LungPoint Virtual Bronchoscopic Navigation (VBN) System
Brief Title: Evaluation of the LungPoint Virtual Bronchoscopic Navigation (VBN) System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Broncus Technologies (Industry)
Collaborators: Heidelberg University (Other)
Responsible Party: Prof. Dr. med Felix Herth, Chief Pneumology and Respiratory Care Medicine, Thoraxklinik, University of Heidelberg
Other Study IDs: Protocol 35
Record Dates: First submitted 2010-01-29; First posted 2010-02-12 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2010-02

CONDITIONS: Lung Neoplasm
Keywords: navigation; bronchoscopy; lymphadenopathy
MeSH Terms: conditions — Lung Neoplasms; Lymphadenopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bronchoscopy, lung neoplasm: Patients who have been recommended for bronchoscopy for the purpose of obtaining a biopsy sample of a central or peripheral pulmonary lesion, diagnosing mediastinal or hilar lymphadenopathy or for lung fiducial placement.
  Interventions: Device: LungPoint Virtual Bronchoscopic Navigation (computer-assisted image-guided bronchoscopic navigation)

INTERVENTIONS:
Device: LungPoint Virtual Bronchoscopic Navigation (computer-assisted image-guided bronchoscopic navigation) — LungPoint Virtual Bronchoscopic Navigation is a product that displays images and information to aid bronchoscopists in guiding the bronchoscope and other instruments to a target location in the lung airways.
  Other Names: LungPoint Virtual Bronchoscopic Navigation

SUMMARY:
To evaluate the role of the LungPoint VBN System in the bronchoscopic access to a target location.

The evaluation will explore:

* Ability of the system to guide a user to one or more target site(s)
* Ease of use of the system (assessment of the user interface)
* Incremental value brought by the use of the system to the successful completion of a case.

DETAILED DESCRIPTION:
Multi-center, prospective, single-arm study. The Study will take the form of a User Evaluation. The Evaluation will require the user to perform several standardized functions (e.g. peripheral lesion sampling, lymph node sampling). In addition, users will be asked about other potential techniques that fall within the intended use of the device.

The evaluation will be conducted in patients who are indicated for procedures that fall within the intended use of the device. Examples of such patients include:

* Patients who have been recommended for bronchoscopy for the purpose of obtaining a biopsy sample of a central or peripheral pulmonary lesion.
* Patients who have been recommended for bronchoscopy for the purpose of diagnosing mediastinal or hilar lymphadenopathy.
* Patients who have been recommended for bronchoscopy for the purpose of lung fiducial placement.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided Informed Consent
* Subject is scheduled for bronchoscopy for the purpose of diagnosing: a central or peripheral pulmonary nodule or mass, infiltrative disease, mediastinal or hilar lymphadenopathy, or placing fiducial markers.
* Subject has a CT scan that is consistent with high-resolution specifications

Exclusion Criteria:

* Patients less than 18 years of age.
* Any patient that the Investigator feels is not appropriate for this study for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in patients who are indicated for procedures that fall within the intended use of the device. Examples of those patient populations are:
  * Patients who have been recommended for bronchoscopy for the purpose of obtaining a biopsy sample of a central or peripheral pulmonary lesion.
  * Patients who have been recommended for bronchoscopy for the purpose of diagnosing mediastinal or hilar lymphadenopathy.
  * Patients who have been recommended for bronchoscopy for the purpose of lung fiducial placement.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-01 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Evidence that LungPoint VBN has a clear role in targeted bronchoscopic procedures | Immediate post-operative (day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Felix Herth, MD, PhD, FCCP, Principal Investigator — Heidelberg University
Locations (1):
- Thoraxklinik, Heidelberg, Germany

REFERENCES:
- [Derived] Eberhardt R, Kahn N, Gompelmann D, Schumann M, Heussel CP, Herth FJ. LungPoint--a new approach to peripheral lesions. J Thorac Oncol. 2010 Oct;5(10):1559-63. doi: 10.1097/JTO.0b013e3181e8b308. PMID 20802352